CLINICAL TRIAL: NCT06770205
Title: Effects of Kendall Exercises Versus Proprioceptive Neuromuscular Facilitation Technique on Pain, Range of Motion, Disability, Craniovertebral and Thoracic Angle in Patients With Upper Cross Syndrome
Brief Title: Kendall Exercises Versus Proprioceptive Neuromuscular Facilitation Technique in Patients With Upper Cross Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0108
Record Dates: First submitted 2024-12-12; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Upper Extremity Dysfunction
Keywords: Pain; Disability; Range of Motion; Craniovertebral angle; Thoracic angle.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial will be conducted at Riphah Clinic Lahore, Sehat medical complex hospital Lahore through consecutive sampling technique on 52 patients which will be allocated using computer generated sampling (random number table) into Group A and Group B. Group A will be treated with kendall exercises and Group B will be treated with Proprioceptive Neuromuscular Facilitation techniques with the frequency that Stretching exercises will be performed actively for 30 second hold and 3 repetitions. Strengthening exercise will be performed for 10 second hold and 10 repetitions. All Exercises will be performed 3 times per week for total of 4 weeks. Outcome measures will be conducted through pain, range of motion, disability craniovertebral and thoracic angle after 4 weeks. Data will be analyzed during SPSS software version 25. The normality of data will be assessed by Shapiro-Wilk test after which it will be decided either parametric or non-parametric test will be used within a g
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physical therapy (Active Comparator): Hot pack and TENS for 10 minutes and massage that will as 3 sessions per week for 4 weeks.
  Interventions: Other: traditional physical therapy
- kendall Exercise Group A (Experimental): The Kendall exercise group participated in 5 sets of consisting of 12 repetitions of postures, each taking 30 seconds, based on Kendall exercise. The Kendall exercise methods were as follows:
  1. Strengthening the deep cervical flexors, lying flat on the back with the chin down and then lifting the head and holding this position for 2-8 seconds to strengthen deep cervical flexors
  2. Stretching the cervical extensors, placing both hands on the occipital area in a sitting position followed by a flexed neck posture with the head down to stretch the cervical extensors
  3. strengthening shoulder retraction, putting a Thera Band around a secure object and pulling the band back with both hands as far as possible to move the shoulder blades toward each other in a standing position
  4. stretching the pectoralis muscle, placing both hands on the occipital area and pulling the elbows back up
  Interventions: Other: kendall Exercise Group A

INTERVENTIONS:
Other: traditional physical therapy — hot pack and TENS for 10 minutes and massage that will as 3 sessions per week for 4 weeks.
  Arms: traditional physical therapy
Other: kendall Exercise Group A — The group B will receive Proprioceptive Neuromuscular Facilitation technique for stretching and rhythmic stabilization technique for strengthening. Proprioceptive Neuromuscular Facilitation (PNF) is a stretching technique utilized to improve muscle elasticity and has been shown to have a positive effect on active and passive range of motions. The PNF group performed the intervention for 30 minutes a day, six times a week, a total of 24 times. (13) In this group, two types of PNF techniques were given:
  1. first is strengthening technique included rhythmic stabilization that is characterized by alternating isometric contractions against resistance, no motion intended to apply for the weak muscles of upper cross syndrome included deep neck flexors specifically lower trapezius and serratus anterior.
  2. Second is stretching technique included contract relax that is resisted isotonic contractions of the restricting muscles (antagonists) followed by relaxation and movement
  Arms: kendall Exercise Group A

SUMMARY:
Upper Crossed Syndrome (UCS) is a postural disorder characterized by a distinct pattern of muscle imbalances within the musculature of the shoulder girdle and cervico-thoracic region. The use of different corrective exercise approaches enhances and improves muscle balance and motor control thereby reducing postural abnormalities. Therefore, the aim of study will be to compare the effects of Kendall exercises versus proprioceptive neuromuscular facilitation technique on pain, range of motion, disability craniovertebral and thoracic angle in patients with upper cross syndrome.

A Randomized Clinical Trial will be conducted at Riphah Clinic Lahore, Sehat medical complex hospital Lahore through consecutive sampling technique on 52 patients which will be allocated using computer generated sampling (random number table) into Group A and Group B. Group A will be treated with kendall exercises and Group B will be treated with Proprioceptive Neuromuscular Facilitation techniques with the frequency that Stretching exercises will be performed actively for 30 second hold and 3 repetitions. Strengthening exercise will be performed for 10 second hold and 10 repetitions. All Exercises will be performed 3 times per week for total of 4 weeks. Outcome measures will be conducted through pain, range of motion, disability craniovertebral and thoracic angle after 4 weeks. Data will be analyzed during SPSS software version 25.

DETAILED DESCRIPTION:
Upper Crossed Syndrome (UCS) is a postural disorder characterized by a distinct pattern of muscle imbalances within the musculature of the shoulder girdle and cervico-thoracic region. This syndrome is typified by tightness and over-facilitation of muscles such as the levator scapulae, pectoralis major, and upper trapezius, juxtaposed with the weakness or inhibition of the serratus anterior, deep neck flexors (specifically scalene), middle trapezius, lower trapezius, and rhomboids. Individuals with UCS typically exhibit a forward head posture, rounded upper back (thoracic kyphosis), elevated and protracted shoulders, and scapular winging. Prolonged and repetitive activities, such as manual material handling, especially when performed in inappropriate postures, can exacerbate the symptoms of UCS. A study involving medical students at the University of Lahore highlighted a concerning prevalence of UCS, with 48.7% of the student population reporting neck pain. The use of different corrective exercise approaches enhances and improves muscle balance and motor control thereby reducing postural abnormalities. Therefore, the aim of study will be to compare the effects of Kendall exercises versus proprioceptive neuromuscular facilitation technique on pain, range of motion, disability craniovertebral and thoracic angle in patients with upper cross syndrome.

A Randomized Clinical Trial will be conducted at Riphah Clinic Lahore, Sehat medical complex hospital Lahore through consecutive sampling technique on 52 patients which will be allocated using computer generated sampling (random number table) into Group A and Group B. Group A will be treated with kendall exercises and Group B will be treated with Proprioceptive Neuromuscular Facilitation techniques with the frequency that Stretching exercises will be performed actively for 30 second hold and 3 repetitions. Strengthening exercise will be performed for 10 second hold and 10 repetitions. All Exercises will be performed 3 times per week for total of 4 weeks. Outcome measures will be conducted through pain, range of motion, disability craniovertebral and thoracic angle after 4 weeks. Data will be analyzed during SPSS software version 25. The normality of data will be assessed by Shapiro-Wilk test after which it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria

* Patients diagnose with upper crossed syndrome.
* To diagnose upper cross syndrome, janda classification or approach will be use. Janda believed that muscle tightness or spasticity is predominant. Often weakness from muscle imbalance results from reciprocal inhibition of the tight antagonist. These patterns lead to postural changes and joint dysfunction and degeneration (23)
* Both genders male and female.
* Participants with constantly or frequently occurring neck-shoulder pain more than 1 month.
* Age between 25 and 50 years (3)
* Pain and restricted range of motion
* NPRS score greater than 3
* Craniovertebral angle < 51 degree. (20)

Exclusion Criteria:

* Tumors
* Pregnancy
* Diagnosed psychological disorders
* Surgery
* Cancer and neuropathies past one year
* Rheumatoid arthritis and cervical instability.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rate scale | 4th day
  Numeric pain rate scale, Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicate worst pain. The NPRS has a validity of (r=0.79-0.96) and a reliability of 0.86-0.89. (16) It takes less than one minute to complete, and can be understood in any language; i.e. there is no language barrier. It is a valid and reliable scale that measures pain intensity and experience.
Neck Disability index | 4th day
  Neck Disability index (NDI), this questionnaire will be used to assess disability. It comprises of 10 items; 7 related to daily living activities, 2 related to pain and 1 related to concentration. Each item is scored from 0 to 5. Total score is expressed as a percentage, with higher scores related to greater disability.

SECONDARY OUTCOMES:
Range of motion | 4th day
  Universal Goniometer (UG) It will measure range of motion of neck in each direction. (19) Universal goniometer is commonly used as a standard method to evaluate joint range of motion as a part of joint assessment.
Craniovertebral angle | 4th day
  APECS/ J-App, This is software will use to measure craniovertebral angle, Craniovertebral angle is measured by taking 2 lateral photographs of the subject in a relaxed seated position without a back support. Spinous process of C7 and the tragus of ear are marked with a body marker. A horizontal line is drawn passing through C7 making a right angle with the vertical. Then, the angle between the line connecting C7 spinous process with the tragus of the ear and the horizontal line, is measured using Image J Software.
Thoracic angle | 4th day
  Flexicurve method using inclinometer, It will use to measure thoracic kyphosis angle.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehab Training and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No